CLINICAL TRIAL: NCT00739180
Title: Physical Activity in Youth: Implications for Reversing Risk Factors for Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Principal Investigator, SoJung Lee, Assistant Professor of Pediatrics, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7-08-JF-27
Record Dates: First submitted 2008-08-20; First posted 2008-08-21 (Estimated); Last update posted 2012-11-06 (Estimated); Status verified 2012-10

CONDITIONS: Abdominal Obesity
Keywords: Childhood obesity; Abdominal obesity; Visceral fat; Insulin resistance; Liver fat; Skeletal muscle lipid; Fitness
MeSH Terms: conditions — Obesity, Abdominal; Pediatric Obesity; Insulin Resistance; Fatty Liver | interventions — Resistance Training; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (Other): Standard care control
  Interventions: Other: Control
- Aerobic Exercise (Active Comparator)
  Interventions: Other: Aerobic exercise
- Resistance Exercise (Active Comparator)
  Interventions: Other: Resistance Exercise

INTERVENTIONS:
Other: Control — Standard care control (no exercise)
  Arms: Control
Other: Resistance Exercise — Supervised resistance exercise using stack weight equipments.
  Arms: Resistance Exercise
Other: Aerobic exercise — Supervised aerobic exercise using treadmills, bikes, and ellipticals
  Arms: Aerobic Exercise

SUMMARY:
In this randomized controlled trial, we will examine the effect of a 3-month exercise training (aerobic exercise versus resistance exercise) without calorie restriction on total and regional adiposity, and risk of type 2 diabetes in overweight children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Healthy overweight (BMI >-95th) youth between 12 and 18 years of age
* Waist circumference >-75th percentile
* Sedentary (no structured exercise >2 times/week for past 6 months)
* Non-smokers, non-diabetic, no medical conditions
* Weight stable for past 3 months

Exclusion Criteria:

* Smokers,
* diabetic,
* psychiatric disorders,
* syndromatic obesity

Ages: 12 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2007-11; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Abdominal obesity, visceral fat | 3 month

SECONDARY OUTCOMES:
Insulin sensitivity and secretion, glucose tolerance | 3 month

CONTACTS AND LOCATIONS:
Overall Officials: SoJung Lee, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh, University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Yu WW, Lee S, Arslanian S, Tamim H, Kuk JL. Effects of Exercise on Resting Metabolic Rate in Adolescents with Overweight and Obesity. Child Obes. 2021 Jun;17(4):249-256. doi: 10.1089/chi.2020.0280. Epub 2021 Mar 18. PMID 33739874
- [Derived] Kuk JL, Lee S. Assessing the utility of cardiorespiratory fitness, visceral fat, and liver fat in predicting changes in insulin sensitivity beyond simple changes in body weight after exercise training in adolescents. Appl Physiol Nutr Metab. 2021 Jan;46(1):55-62. doi: 10.1139/apnm-2020-0284. Epub 2020 Jul 16. PMID 32674604
- [Derived] Kuk JL, Lee S. Sex and Ethnic Differences in the Relationship between Changes in Anthropometric Measurements and Visceral Fat in Adolescents with Obesity. J Pediatr. 2019 Oct;213:121-127. doi: 10.1016/j.jpeds.2019.05.052. Epub 2019 Jun 22. PMID 31235380